CLINICAL TRIAL: NCT07253480
Title: Correlation of Diaphragm Shear-Wave Elastography With Transdiaphragmatic Pressure in Healthy Adults: a Feasibility Study
Acronym: PLEASSURE 1
Status: Not yet recruiting | Type: Observational
Sponsor: Isala (Other)
Collaborators: University Medical Center Groningen (Other)
Responsible Party: Principal Investigator, Wytze de Boer, Principal investigator, University Medical Center Groningen
Other Study IDs: PLEASSURE 1
Record Dates: First submitted 2025-11-19; First posted 2025-11-28 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Diaphragm Ultrasound; Diaphragm Dysfunction; Health Adult Subjects
Keywords: diaphragm; ultrasound; diaphragmatic pressure; shear-wave elastography

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- healthy adults: prospective validation cohort of healthy adults
  Interventions: Diagnostic Test: shear wave elastography of the diaphragm

INTERVENTIONS:
Diagnostic Test: shear wave elastography of the diaphragm — Participants will undergo simultaneous measurements of diaphragm SWE, transdiaphragmatic pressure (Pdi = Pga-Pes), and inspiratory mouth pressures (Pmo) at rest and during inspiratory efforts at 20%, 40%, and 60% of PImax. SWE will be performed twice by different operators to assess inter-rater reliability. The primary analysis will determine within-individual and overall correlations between SWE and Pdi.
  - Pearson correlation coefficient repeated-measures correlation coefficient between SWE and Pdi across inspiratory efforts.

SUMMARY:
Changes in intrapleural pressure after lung volume reduction in Chronic Obstructive Pulmonary disease (COPD) patients can lead to complications, including an increased risk of pneumothorax. This procedure, intended to improve lung function, may disturb the pressure balance within the pleural space, potentially precipitating pneumothorax. Careful monitoring of intrapleural pressure could help predict patients at risk. However, intrapleural pressure can currently only be measured invasively. Diaphragm shear-wave elastography (SWE) has been shown to reflect transdiaphragmatic pressure during isovolumetric inspiratory efforts and ventilation against inspiratory loading, and therefore may serve as a non-invasive surrogate for intrapleural pressure. This project outlines a stepwise study plan to evaluate SWE as a tool for intrapleural pressure monitoring (Figure 1). The project only moves to the next phase is the study previous phase was achieved successfully. The current protocol involves the first phase: to validate diaphragm SWE against transdiaphragmatic pressure and assess measurement reliability for local ultrasound systems in healthy adults.This prospective, single-centre, observational validation study will include twelve healthy adult volunteers. During a single study session, participants will perform standardized inspiratory efforts while simultaneous measurements of diaphragm SWE, transdiaphragmatic pressure (via esophageal and gastric balloon catheters), and mouth pressures are obtained. These methods are routinely applied in physiological research and carry minimal risk. Apart from brief nasal or throat discomfort during catheter placement, no significant adverse effects are expected. By establishing the relationship between diaphragm SWE, transdiaphragmatic pressure, and mouth pressures, this study aims to provide the essential validation step for future clinical research in COPD patients following lung volume reduction.

DETAILED DESCRIPTION:
Rationale:

Changes in intrapleural pressure after lung volume reduction in COPD patients may contribute to pneumothorax. Non-invasive monitoring of pleural pressure could help identify patients at risk. Diaphragm shear-wave elastography (SWE) has shown potential to reflect transdiaphragmatic pressure (Pdi), but has not yet been validated across ultrasound systems. This study aims to validate diaphragm SWE against gold-standard Pdi and mouth pressures in healthy volunteers before applying the technique in COPD patients.

Objective:

To validate diaphragm SWE as a non-invasive measure of inspiratory effort by assessing its correlation with transdiaphragmatic pressure (Pdi) and mouth pressure (PImax and submaximal inspiratory pressures). Secondary objectives are to determine feasibility and inter-rater reliability of SWE measurements.

Study design:

Prospective, single-centre, observational validation study.

Study population:

Twelve healthy adults aged 18-60 years, BMI 18-30 kg/m², without respiratory, neuromuscular or cardiothoracic disease.

Main study parameters/endpoints:

Participants will undergo simultaneous measurements of diaphragm SWE, transdiaphragmatic pressure (Pdi = Pga-Pes), and inspiratory mouth pressures (Pmo) at rest and during inspiratory efforts at 20%, 40%, and 60% of PImax. SWE will be performed twice by different operators to assess inter-rater reliability. The primary analysis will determine within-individual and overall correlations between SWE and Pdi.

- Pearson correlation coefficient repeated-measures correlation coefficient between SWE and Pdi across inspiratory efforts.

Nature and extent of the burden and risks associated with participation, benefit and group relatedness:

The study involves a single measurement session (~1-2 hours). Procedures include nasal insertion of esophageal and gastric balloon catheters, mouth pressure measurements, and diaphragm ultrasound. These are routinely used physiological techniques with mild, transient, discomfort (e.g., mild throat or nasal irritation). No therapeutic intervention or follow-up is required. Risks are considered negligible and proportionate to the scientific value of the validation.

ELIGIBILITY:
Inclusion Criteria:

* 18-60 years, BMI 18-30 kg/m²
* No known respiratory, neuromuscular, or cardiothoracic disease
* Able to perform inspiratory maneuvers and consent.

Exclusion Criteria:

* Pregnancy
* History of smoking (> 10 pack years)
* Impaired swallowing, as well as esophageal diseases, or disorders at the level of the gastroesophageal sphincter

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Healthy adults.
Sampling Method: Probability Sample
Enrollment: 12 (Estimated)
Dates: Start 2026-04 (Estimated); Primary Completion 2026-06 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
- Pearson correlation coefficient repeated-measures correlation coefficient between SWE and Pdi across inspiratory efforts. | 1 hour
  Participants will undergo simultaneous measurements of diaphragm SWE, transdiaphragmatic pressure (Pdi = Pga-Pes), and inspiratory mouth pressures (Pmo) at rest and during inspiratory efforts at 20%, 40%, and 60% of PImax. SWE will be performed twice by different operators to assess inter-rater reliability. The primary analysis will determine within-individual and overall correlations between SWE and Pdi.

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Centre Groningen, Groningen, Provincie Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided
small feasibility study